CLINICAL TRIAL: NCT05674084
Title: Influence of Vasopressor Support and Mean Arterial Pressure on Capillary Refill Time Values in Critically Ill Patients: Prospective, Observational Study
Brief Title: Vasopressor Support, Mean Arterial Pressure and Capillary Refill Time in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Łukasz Krzych, Professor, Medical University of Silesia
Other Study IDs: PCN/CBN/0052/KB/242/22
Record Dates: First submitted 2022-12-11; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Critical Illness
Keywords: capillary refill time; norepinephrine; epinephrine; argipressin; dobutamine; mean arterial pressure
MeSH Terms: conditions — Critical Illness; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Critically ill patients undergoing any vasopressor treatment. CRT will be measured over the course of hospitalization. Maximal number of CRT measurements from a single patient is limited to 5.
  Interventions: Diagnostic Test: Capillary refill time

INTERVENTIONS:
Diagnostic Test: Capillary refill time — CRT will be measured by applying firm pressure to the ventral surface of the index finger distal phalanx with a glass microscope slide. The pressure will be increased until the skin is blank and then maintained for 10 seconds. The time for return of the normal skin color will be registered with a chronometer, and > 3 seconds is defined as abnormal. Light and ambient temperature will be the same for all individuals.

SUMMARY:
The goal of this observational study is to learn whether different doses of various vasopressor drugs influence capillary refill time (CRT) value in crtically ill patients. The main questions it aims to answer are:

* How do vasopressor drugs determine CRT value
* How does mean arterial pressure (MAP) determine CRT value
* How often CRT value is normal (< 3 sec) despite hypotensive MAP (<65 mmHg)

Participants will have the CRT measured over the course of the ICU hospitalization. At the end of the study, multiple linear regression will be performed to verify whether different doses of vasopressor drugs influence CRT value.

DETAILED DESCRIPTION:
The goal of this observational study is to learn whether different doses of various vasopressor drugs influence capillary refill time (CRT) value in critically ill patients. The main questions it aims to answer are:

* How does norepinephrine dose influence CRT value
* How does epinephrine dose influence CRT value
* How does argipressin dose influence CRT value
* How does dobutamine dose influence CRT value
* How does mean arterial pressure (MAP) determine CRT value
* How often CRT value is normal (< 3 sec) despite hypotensive MAP (<65 mmHg)

Participants will have the CRT measured over the course of the ICU hospitalization. At the end of the study, multiple linear regression will be performed to verify whether different doses of vasopressor drugs influence CRT value. CRT will be a dependent variable. Independent variables will be as follows: age, MAP, norepinephrine dose, epinephrine dose, argipressin dose, dobutamine dose.

CRT measurements will be performed in a standarized rigor (light, chronometer, pressure and ambient temperature will be the same in all patients)

ELIGIBILITY:
Inclusion Criteria:

* critical illness requiring vasopressor support
* invasive blood pressure monitoring

Exclusion Criteria:

* finger distal phalanx not available
* patient in a room of suboptimal ambient temperature

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients requiring vasopressor support will be included in the study. Over the course of the ICU hospitalization, a maximal number of 5 CRT measurements will be made.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of norepinephrine dose on CRT value | Through study completion, an average of 1 year
  In a multiple linear regression, it will be verified whether different doses of norepinephrine determine CRT value.
Effect of mean arterial pressure on CRT value | Through study completion, an average of 1 year
  In a multiple linear regression, it will be verified whether different values of MAP determine CRT value.

SECONDARY OUTCOMES:
Effect of epinephrine dose on CRT value | Through study completion, an average of 1 year
  In a multiple linear regression, it will be verified whether different doses of epinephrine determine CRT value.
Effect of argipressin dose on CRT value | Through study completion, an average of 1 year
  In a multiple linear regression, it will be verified whether different doses of argipressin determine CRT value.
Effect of dobutamine dose on CRT value | Through study completion, an average of 1 year
  In a multiple linear regression, it will be verified whether different doses of dobutamine determine CRT value.
CRT value in MAP <65 mmHg | Through study completion, an average of 1 year
  It will be analyzed whether in hypotensive conditions (MAP <65 mmHg), CRT values are normal (< 3 sec)

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Krzych, Professor, Study Chair — Medical University of Silesia
Locations (1):
- University Clinical Center named after prof. K. Gibiński of the Medical University of Silesia in Katowice, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire D, Gotlib A, King J. Capillary Refill Time. 2023 Apr 23. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557753/ PMID 32491685
- [Background] Hernandez G, Ospina-Tascon GA, Damiani LP, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Granda-Luna V, Cavalcanti AB, Bakker J; The ANDROMEDA SHOCK Investigators and the Latin America Intensive Care Network (LIVEN); Hernandez G, Ospina-Tascon G, Petri Damiani L, Estenssoro E, Dubin A, Hurtado J, Friedman G, Castro R, Alegria L, Teboul JL, Cecconi M, Cecconi M, Ferri G, Jibaja M, Pairumani R, Fernandez P, Barahona D, Cavalcanti AB, Bakker J, Hernandez G, Alegria L, Ferri G, Rodriguez N, Holger P, Soto N, Pozo M, Bakker J, Cook D, Vincent JL, Rhodes A, Kavanagh BP, Dellinger P, Rietdijk W, Carpio D, Pavez N, Henriquez E, Bravo S, Valenzuela ED, Vera M, Dreyse J, Oviedo V, Cid MA, Larroulet M, Petruska E, Sarabia C, Gallardo D, Sanchez JE, Gonzalez H, Arancibia JM, Munoz A, Ramirez G, Aravena F, Aquevedo A, Zambrano F, Bozinovic M, Valle F, Ramirez M, Rossel V, Munoz P, Ceballos C, Esveile C, Carmona C, Candia E, Mendoza D, Sanchez A, Ponce D, Ponce D, Lastra J, Nahuelpan B, Fasce F, Luengo C, Medel N, Cortes C, Campassi L, Rubatto P, Horna N, Furche M, Pendino JC, Bettini L, Lovesio C, Gonzalez MC, Rodruguez J, Canales H, Caminos F, Galletti C, Minoldo E, Aramburu MJ, Olmos D, Nin N, Tenzi J, Quiroga C, Lacuesta P, Gaudin A, Pais R, Silvestre A, Olivera G, Rieppi G, Berrutti D, Ochoa M, Cobos P, Vintimilla F, Ramirez V, Tobar M, Garcia F, Picoita F, Remache N, Granda V, Paredes F, Barzallo E, Garces P, Guerrero F, Salazar S, Torres G, Tana C, Calahorrano J, Solis F, Torres P, Herrera L, Ornes A, Perez V, Delgado G, Lopez A, Espinosa E, Moreira J, Salcedo B, Villacres I, Suing J, Lopez M, Gomez L, Toctaquiza G, Cadena Zapata M, Orazabal MA, Pardo Espejo R, Jimenez J, Calderon A, Paredes G, Barberan JL, Moya T, Atehortua H, Sabogal R, Ortiz G, Lara A, Sanchez F, Hernan Portilla A, Davila H, Mora JA, Calderon LE, Alvarez I, Escobar E, Bejarano A, Bustamante LA, Aldana JL. Effect of a Resuscitation Strategy Targeting Peripheral Perfusion Status vs Serum Lactate Levels on 28-Day Mortality Among Patients With Septic Shock: The ANDROMEDA-SHOCK Randomized Clinical Trial. JAMA. 2019 Feb 19;321(7):654-664. doi: 10.1001/jama.2019.0071. PMID 30772908
- [Background] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770
- [Background] Dubin A, Pozo MO, Casabella CA, Palizas F Jr, Murias G, Moseinco MC, Kanoore Edul VS, Palizas F, Estenssoro E, Ince C. Increasing arterial blood pressure with norepinephrine does not improve microcirculatory blood flow: a prospective study. Crit Care. 2009;13(3):R92. doi: 10.1186/cc7922. Epub 2009 Jun 17. PMID 19534818